CLINICAL TRIAL: NCT06504342
Title: Pilot Trial of Time Restricted Eating to Support an Adaptive Innovative Clinical Trial of Combined Chronotherapies for Mania in Bipolar Disorder
Brief Title: Clocks in Sync - Circadian Rhythm and Bipolar Mania
Acronym: CIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 20240219-01H
Record Dates: First submitted 2024-06-25; First posted 2024-07-16 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Bipolar Disorder; Mania
Keywords: Chronotherapy; Blue-blocking glasses; Time-restricted eating
MeSH Terms: conditions — Bipolar Disorder; Mania; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: 2 by 2 factorial design. Only 3 of the 4 arms will be implemented, with the double control arm not implemented in the pilot.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The time-restricted eating intervention will be single-blind, only the investigators/outcomes assessors will be blinded. The tinted glasses intervention will be double-blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Blue-blocking glasses and time-restricted eating (Experimental): Participants will be wearing the experimental blue-blocking glasses and follow time-restricted eating from 6pm-8am.
  Interventions: Device: Blue-blocking glasses; Behavioral: Time-restricted eating
- Blue-blocking glasses and no time-restricted eating (Active Comparator): Participants will only be wearing the experimental blue-blocking glasses from 6pm-8am.
  Interventions: Device: Blue-blocking glasses
- Lightly tinted glasses and time-restricted eating (Active Comparator): Participants will be wearing the control lightly tinted glasses and follow time-restricted eating from 6pm-8am.
  Interventions: Behavioral: Time-restricted eating; Device: Lightly tinted glasses

INTERVENTIONS:
Device: Blue-blocking glasses — These lenses will filter ~10% of visible light across the visible light range (including in the range activating melanopsin) with complete blockade of ultraviolet light.
  Arms: Blue-blocking glasses and no time-restricted eating; Blue-blocking glasses and time-restricted eating
Behavioral: Time-restricted eating — Avoid caloric food intake for a fourteen-hour period overnight from 6 p.m. to 8 a.m
  Arms: Blue-blocking glasses and time-restricted eating; Lightly tinted glasses and time-restricted eating
Device: Lightly tinted glasses — These lenses block shorter wavelengths of light, mainly ultraviolet light.
  Arms: Lightly tinted glasses and time-restricted eating

SUMMARY:
The sleep-wake cycle is severely disrupted during an episode of mania. Often mania is treated with medications that can come with significant side effects. Years of patient and family engagement with this population have revealed great interest in therapies targeting the sleep-wake cycle. However, there is still a lack of studies to support using these treatments for mania. Patient partners are especially interested in two specific therapies for mania, blue-blocking glasses and time-restricted eating, because of their perceived feasibility and safety. This pilot study will formally investigate the feasibility and effectiveness of these therapies for participants with mania, an understudied population that faces many difficulties even after recovery. The pilot study will collect interviews to identify barriers and ways to better support patients with mania using the therapies. The study will also investigate how well these therapies can treat manic symptoms and restore sleep-wake cycles by tracking symptom rating scales and measuring activity levels. Results from this pilot will be used to direct a larger study that will use a state-of-the art design to test the effectiveness of both therapies alone and in combination.

DETAILED DESCRIPTION:
This pilot study will assess feasibility and preliminary data for a novel circadian intervention in a clinical population that has been understudied, patients dealing with manic episodes of bipolar disorder, with an equity, diversity, and inclusion plan to ensure broad demographic representation.

The investigators' long-term goal is to conduct an innovative adaptive, 2x2 factorial study of these two interventions to determine the effects of each individual component and potential synergistic interactions. An adaptive design will allow interim analyses for sample size during which futility can also be assessed. This may potentially reduce cost and time of the later full trial, while ensuring that relevant findings are obtained. To inform a later 2x2 factorial study, researchers will need to gather data on the feasibility of time restricted eating in mania and identify any forms of support required to facilitate this chronotherapy. This is a randomized, parallel three group pilot study of blue-blocking glasses, time restricted eating, or blue-blocking glasses plus time-restricted eating in inpatients with mania. This project has three specific aims:

Aim 1: To assess the feasibility of time restricted eating (10:14 of diurnal eating to nocturnal fasting based on patient partners' input) as an adjunctive treatment for mania in an inpatient setting. Feasibility will be assessed through monitoring of adherence and qualitative semi-structured interviews with patient participants when they exit the study and staff near the study end date. The purpose of these interviews is to identify any challenges or barriers in implementing this treatment, alone or in combination with blue blocking glasses, and what supports might be needed. The research team will also assess willingness to participate in the study through assessment of participation rates and reasons for accepting or declining.

Aim 2: The investigators will secondarily compare differences between groups on the Young Mania Rating Scale (YMRS), which will be the primary outcome for the future trial.

Aim 3 (exploratory): To explore changes in measures of circadian rhythms and sleep, including as measured with actigraphy and other non-invasive monitoring measures, with the interventions and in relation to recovery from mania.

ELIGIBILITY:
Inclusion Criteria:

* Be over age 16
* Have DSM-5-defined manic symptoms that persist beyond the physiological effects of a substance and a YMRS≥20
* Be willing to have investigators obtain information from the treatment team and electronic medical record
* Participants must be able to read and understand English or French.
* Be willing and able to provide informed consent.

Exclusion Criteria:

* Have a history of eating disorders.
* Have a diagnosis of moderate to severe traumatic brain injury with residual or long-term effects, parenchymal brain surgery or stroke
* Have a neurocognitive disorder
* Take hypoglycemia-inducing medications
* Be pregnant/lactating women
* Have a diagnosis of sleep apnea
* Have any other medical condition for which physician or investigator team expresses concern about safety or ability to participate in the study.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-09-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Time-Restricted Eating: 1) Study Participation | Over the lifetime of the study starting at the first patient approached until recruitment is stopped.
  Feasibility of time restricted eating for inpatients with mania as assessed by study participation, defined as the ratio of patients who consent to participate in the study after being approached by the research team. This will be reported as a ratio with the number of participants who consented as the numerator and the total number of patients approached for participation in the study as the denominator.
Feasibility of Time-Restricted Eating: 2) Adherence to Protocol | Baseline to Week 2 or until discharge, whichever comes first
  Feasibility of time restricted eating for inpatients with mania as assessed by self-reported and observed adherence. At each study visit, the research team will consider the participants' self-report, notes in the medical record, and their own observations to select a rating on a Likert scale indicating how closely the participant has adhered to the schedule of their assigned intervention(s): a) Fully adherent; b) Almost fully adherent; c) Mostly adherent; d) Half adherent; e) Mostly non-adherent; f) Barely adherent; g) Not adherent.
Feasibility of Time-Restricted Eating: 3) Qualitative Interviews | One interview prior to the participant's discharge, at the end of their participation in the study.
  Feasibility of time restricted eating for inpatients with mania as assessed by qualitative semi-structured interview. The research team will conduct a semi-structured interview with participants to elicit their perspective on the feasibility of time restricted eating in the context of an inpatient research study.

SECONDARY OUTCOMES:
Change in the Young Mania Rating Scale | Baseline to Week 2 or until discharge, whichever comes first
  The Young Mania Rating Scale is used to evaluate the severity of manic symptoms at baseline and over time in individuals with mania. It is an 11-item scale and total score ranges from 0 to 60 where higher scores indicate more severe mania, thus, a negative change (or decrease) from baseline indicates a reduction (or improvement) in manic symptoms. Total score ≤12 indicates remission (13-19=minimal symptoms; 20-25=mild mania, 26-37=moderate mania, 38-60=severe mania).
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score | Baseline to Week 2 or until discharge, whichever comes first
  The Montgomery-Åsberg Depression Rating Scale is a clinician-rated depression scale used to assess depression symptom severity. It consists of 10 scored items, each scaled from 0 to 6 and the entire form totaling 0 to 60. The higher the score, the more severe the symptoms. A total score of 0-8 = remission/symptoms absent; 9-17 = mild depression; 18-34 = moderate depression; 35-60 = severe depression
Change in the General Anxiety Disorder Questionnaire- 7-Item Measuring Severity of Anxiety Symptoms (GAD-7) | Baseline to Week 2 or until discharge, whichever comes first
  Self-reported measurement of the severity of anxiety symptoms experienced within the last two weeks. It consists of 7 scored items and one follow-up question. Each of the 7 scored items generates a value from 0 (not at all) to 3 (nearly every day), yielding a total score ranging from 0 to 21, with higher scores indicating more severe symptoms of anxiety. These scores are interpreted in the following manner: a score of 0-4 indicates little or no anxiety, a score of 5-9 indicates mild anxiety, a score of 10-14 indicates moderate anxiety, and a score of 15-21 indicates severe anxiety. Generally, a score of 10 or above is considered to be a clinical cutoff implying that the respondent may be suffering from a general anxiety disorder.
Change in The Morning Evening Questionnaire - 19-Item Self-Assessment Questionnaire for Sleep Rhythms, Habits and Fatigue (MEQ) | Baseline; Week 1; Week 2 or until discharge, whichever comes first
  This questionnaire has 19 questions, each with a number of points. Scores can range from 16-86. Scores of 41 and below indicate "evening types." Scores of 59 and above indicate "morning types." Scores between 42-58 indicate "intermediate types."
Change in The Pittsburgh Sleep Quality Index - 18-Item Self-Assessment to Evaluate Sleep Quality (PSQI) | Baseline; Week 1; Week 2 or until discharge, whichever comes first
  The Pittsburg Sleep Quality Index Questionnaire is self-administered questionnaire designed to evaluate sleep quality consisting of 18 items that in turn are comprised of seven components, which include subjective sleep quality, sleep duration, sleep onset, habitual sleep efficiency, sleep disturbances, use of sleeping medications and daytime dysfunction. Each weighted equally on a 0-3 scale to be summed to yield a global PSQI score, which ranges between 0 and 21, where the higher the scores, the worse the sleep quality.
Change in Circadian Rhythms: 1) Actigraphy | One week of continuous wearing starting at the Baseline visit.
  Wrist actigraphy data that captures the participant's activity level and their exposure to ambient light. The participant will wear the device continuously for one week. The research team will compare the data from different days to assess any changes in activity or light exposure.
Change in Circadian Rhythms: 2) Heart Rate | Two 24-hour periods: one starting at the Baseline visit and the other starting at the Week 1 visit.
  Heart rate monitors will be used to capture data from two different 24-hour periods one week apart. The research team will compare the two time periods for each participant to determine if there are changes.
Change in Circadian Rhythms: 3) Body Temperature | Two 24-hour periods: one starting at the Baseline visit and the other starting at the Week 1 visit.
  Body temperature monitoring using a device attached to the skin of the abdomen near the navel. The device will capture temperature data for two 24-hour periods one week apart. The research team will compare the two time periods for each participant to determine if there are changes.

CONTACTS AND LOCATIONS:
Overall Officials: Jess G Fiedorowicz, MD, PHD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Insitute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No